CLINICAL TRIAL: NCT04284930
Title: Prospective, Randomized, Controlled Comparison of Local Anesthetic Infusion Pump Versus DepoFoam Bupivacaine For Pain Management After Unilateral Deep Inferior Epigastic Perforator Free Flap Reconstruction
Brief Title: Comparison of Local Anesthetic Infusion Pump Versus Depofoam Bupivacaine for Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Risal Djohan, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-1535
Record Dates: First submitted 2016-08-12; First posted 2020-02-26 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Pain, Postoperative
Keywords: local anesthetic continuous infusion pump; local injection of Exparel
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Depobupivacaine (Experimental): Group 1 will receive an injection of 166mg of Depobupivacaine diluted in 60 ml.
  Interventions: Drug: Depobupivacaine
- OnQ Pump (Active Comparator): Group 2 : The OnQ group will receive an infiltration via an OnQ soaker catheter of 0.25% bupivacaine at 4 ml/hour.
  Interventions: Drug: OnQ pump
- bupivacaine (Active Comparator): Group 3: The 0.25% bupivacaine patients will receive 2mg/kg of 0.25% bupivacaine.
  Interventions: Drug: 0.25% Bupivacaine

INTERVENTIONS:
Drug: Depobupivacaine — surgeons receive schematic for injection of Depobupivacaine. Subjects receive an injection of 166mg depobupivacaine. Injection on either side of the suture line, injected directly into the fascia.
  Other Names: Exparel
  Arms: Depobupivacaine
Drug: OnQ pump — group 2: Surgeons receive instruction sheet with specific placement of catheter. All patients have two OnQ soaker catheters installed into abdominal donor site before donor closure.
  Arms: OnQ Pump
Drug: 0.25% Bupivacaine — group 3: given 0.25% bupivacaine without epinephrine between internal oblique and transverse abdominal muscle.
  Other Names: Marcaine
  Arms: bupivacaine

SUMMARY:
Effective post surgical pain control in patients undergoing unilateral deep inferior epigastric perforator (DIEP) free flap reconstruction.

DETAILED DESCRIPTION:
Critical to patient recovery, and can contribute to faster patient mobilization, shorter hospital stays and reduced health care costs. The administration of local anesthetics via wound infiltration is standard of care and an effective practice for post surgical pain management, However this method only provides relatively brief analgesia, usually lasting only 12 hours. Other FDA approved delivery systems using an indwelling fusion pump catheter (On-Q pump) are currently being used in our practice and may be used to extend the duration of action of locally administered analgesia by continuously infusing anesthetic into the wound. Alternatively, a depot form of bupivacaine has been FDA approved and currently used to deliver a single dose administered via wound infiltration for prolonged analgesia by allowing for the diffusion of the drug over an extended period of time. Both of these products are used as a standard practice during DIEP free flap reconstructions. However, no studies compare the efficacy of these two methods patients undergong unilateral DIEP flap reconstructions has been done in a prospective, randomized control manner.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant women
* age 18 years or older
* scheduled to have unilateral DIEP flap breast reconstruction.
* Must have ASA physical status classification of 1,2, or 3

Exclusion Criteria:

* concurrent or recent medical condition that could interfere with study participation
* history of any of the following:
* hepatitis
* alcohol/substance abuse
* uncontrolled psychiatric disorders
* known allergy/ contraindication to any of the following:
* amide-type local anesthetics
* opioids
* propofol
* Body weight of less than 50 kg
* have participated in another study involving an investigational medication with in the past 30 days
* taking analgesics, antidepressants, or glucocorticoids within the 3 days before surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Risal Djohan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was closed at interim analysis due to analyzed findings supporting use of exparel for pain control. We felt it would be unethical to continue to with overwhelming positive results.
Period: Overall Study
Arm/Group | Depobupivacaine | OnQ Pump | Bupivacaine
Started | 8 | 5 | 8
Completed | 8 | 5 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Depobupivacaine | OnQ Pump | Bupivacaine | Total
Number analyzed (Participants) | 8 | 5 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (7.1) | 51.33 (6.25) | 50 (5.7) | 51.12 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 8 | 21
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Race white | 8 | 5 | 8 | 21
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Total Narcotic Usage
Description: Post-op pain measured by total post-op Morphine equivalents
Time Frame: total hospital stay, an average of 3 days
Measure: Mean (Standard Deviation); unit: mg/kg/day morphine
Arm/Group | Depobupivacaine | OnQ Pump | Bupivacaine
Number analyzed (Participants) | 8 | 5 | 8
mg/kg/day morphine | 0.8 (0.5) | .13 (.1) | 0.18 (0.1)

ADVERSE EVENTS:
Time Frame: The adverse events are collected while the patients were in the hospital, which was an average of 3 days
Arm/Group | Depobupivacaine | OnQ Pump | Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT04284930/Prot_SAP_000.pdf